CLINICAL TRIAL: NCT03075176
Title: Outcomes of Topography-guided LASIK and Photorefractive Keratectomy Compared to Wavefront Optimized LASIK and Photorefractive Keratectomy
Brief Title: Topo-guided LASIK and Photorefractive Keratectomy vs Wavefront LASIK and Photorefractive Keratectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of the bias in who qualified for the study it became apparent we would not get any statistically valid results.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Mark Mifflin, Professor, Ophthalmology/Visual Sciences, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB # 95434
Record Dates: First submitted 2017-02-18; First posted 2017-03-09 (Actual); Results first posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-06

CONDITIONS: Surgery; Myopia
Keywords: Photorefractive keratectomy; Laser-assisted in situ keratomileusis
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Each participant will receive wavefront optimized surgery in one eye and topography-guided surgery in the second eye.
Who Masked: Participant
Masking Description: Participants will be masked as to which type of surgery they receive in either eye.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Wavefront optimized LASIK (Active Comparator): Participants who chose to have LASIK surgery were assigned to have Wavefront optimized LASIK in one eye and Topography-guided LASIK in the other eye (randomly chosen).
  Interventions: Device: Wavefront optimized LASIK; Device: Topography-guided LASIK
- Wavefront optimized Photorefractive Keratectomy (Active Comparator): Participants who chose to have Photorefractive Keratectomy surgery were assigned to have Wavefront optimized Photorefractive Keratectomy in one eye and Topography-guided Photorefractive Keratectomy in the other eye (randomly chosen).
  Interventions: Device: Wavefront optimized Photorefractive Keratectomy; Device: Topography-guided Photorefractive Keratectomy
- Topography-guided LASIK (Active Comparator): Participants who chose to have LASIK surgery were assigned to have Topography-guided LASIK in one eye and Wavefront optimized LASIK in the other eye (randomly chosen).
  Interventions: Device: Wavefront optimized LASIK; Device: Topography-guided LASIK
- Topography-guided Photorefractive Keratectomy (Active Comparator): Participants who chose to have Photorefractive Keratectomy surgery were assigned to have Topography-guided Photorefractive Keratectomy in one eye and Wavefront optimized Photorefractive Keratectomy in the other eye (randomly chosen).
  Interventions: Device: Wavefront optimized Photorefractive Keratectomy; Device: Topography-guided Photorefractive Keratectomy

INTERVENTIONS:
Device: Wavefront optimized LASIK — Wavefront optimized laser vision correction
  Arms: Topography-guided LASIK; Wavefront optimized LASIK
Device: Wavefront optimized Photorefractive Keratectomy — Wavefront optimized laser vision correction
  Arms: Topography-guided Photorefractive Keratectomy; Wavefront optimized Photorefractive Keratectomy
Device: Topography-guided LASIK — Topography-guided laser vision correction
  Arms: Topography-guided LASIK; Wavefront optimized LASIK
Device: Topography-guided Photorefractive Keratectomy — Topography-guided laser vision correction
  Arms: Topography-guided Photorefractive Keratectomy; Wavefront optimized Photorefractive Keratectomy

SUMMARY:
This study evaluates the difference in results between eyes that have been treated wavefront optimized laser vision correction (either LASIK or Photorefractive Keratectomy) compared to eyes treated with topography-guided laser vision correction (either LASIK or Photorefractive Keratectomy). Each participant will receive wavefront optimized correction in one eye and topography-guided correction in the other.

DETAILED DESCRIPTION:
Participants will have an in depth discussion with our refractive surgery coordinator regarding refractive surgery. Patients will choose LASIK or Photorefractive Keratectomy surgery based on our standard pre-operative discussion that is provided to all patients. As is standard for laser refractive candidates, the advantages and disadvantages of LASIK and Photorefractive Keratectomy compared to the other refractive surgical options will be discussed. Following patient selection of their preferred type of refractive procedure they will be randomized as discussed below, and only patients who elect for LASIK or Photorefractive Keratectomy will be included in our study.

Prior to surgery, one eye from each patient will be randomly assigned to receive either Wavefront optimized or Topography Guided treatment. Each patient in the study will have a fellow eye enrolled in the other treatment group. Patients will either receive LASIK treatment or Photorefractive Keratectomy treatment in both eyes but the eyes will be randomized to topography guided or wavefront optimized forms of treatment.

ELIGIBILITY:
Inclusion Criteria:

* All subjects who are deemed suitable candidates for laser refractive surgery after routine refractive surgery screening will be considered eligible for participation in this study.

Subjects must be at least 21 years of age and not pregnant or nursing (due to fluctuations in visual parameters during pregnancy)

Exclusion Criteria:

* Any patient who is not a suitable candidate for LASIK or PRK will not be included.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mifflin, MD, Principal Investigator — University of Utah Moran Eye Center
Locations (1):
- Moran Eye Center - Midvalley Location, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 39 participants were randomized, one participant withdrew, 38 completed wavefront surgery on one eye and topoguided surgery on the other eye. A total of 76 eyes were treated.
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | Wavefront Optimized LASIK | Wavefront Optimized Photorefractive Keratectomy | Topography-guided LASIK | Topography-guided Photorefractive Keratectomy
Started | 18; 18 eyes (In this section, we are not able to enter the correct value in the Total columns to reflect the number of unique participants. 18 participants underwent LASIK (of which 18 eyes received wavefront optimized treatment and 18 eyes received topography-guided treatment). The format provided in CT.gov automatically double-counts the row of "Participants" via calculation and does not allow us to accurately reflect each person in a "split-person" study.) | 20; 20 eyes (In this section, we are not able to enter the correct value in the Total columns to reflect the number of unique participants. 20 participants underwent PRK (of which 20 eyes received wavefront optimized treatment and 20 eyes received topography-guided treatment). The format provided in CT.gov automatically double-counts the row of "Participants" via calculation and does not allow us to accurately reflect each person in a "split-person" study.) | 18; 18 eyes (In this section, we are not able to enter the correct value in the Total columns to reflect the number of unique participants. 18 participants underwent LASIK (of which 18 eyes received wavefront optimized treatment and 18 eyes received topography-guided treatment). The format provided in CT.gov automatically double-counts the row of "Participants" via calculation and does not allow us to accurately reflect each person in a "split-person" study.) | 20; 20 eyes (In this section, we are not able to enter the correct value in the Total columns to reflect the number of unique participants. 20 participants underwent PRK (of which 20 eyes received wavefront optimized treatment and 20 eyes received topography-guided treatment). The format provided in CT.gov automatically double-counts the row of "Participants" via calculation and does not allow us to accurately reflect each person in a "split-person" study.)
Completed | 18; 18 eyes | 20; 20 eyes | 18; 18 eyes | 20; 20 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Wavefront Optimized LASIK | Wavefront Optimized Photorefractive Keratectomy | Topography-guided LASIK | Topography-guided Photorefractive Keratectomy | Total
Number analyzed (Participants) | 18 | 20 | 18 | 20 | 38
Number analyzed (Eyes) | 18 | 20 | 18 | 20 | 76
Age, Categorical [Count of Units; unit: Eyes]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 20 | 18 | 20 | 76
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Units; unit: Eyes]
  Female | 11 | 10 | 11 | 10 | 42
  Male | 7 | 10 | 7 | 10 | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
    (all) |  |  |  |  | 0
Region of Enrollment [Number; unit: Eyes]
  United States | 18 | 20 | 18 | 20 | 76

OUTCOME MEASURES:

1. Primary Outcome: Change in Uncorrected Visual Acuity From Baseline to Month 12
Description: Uncorrected visual acuity will be tested pre-operatively through month 12
Time Frame: 12 months
Population: Twelve month data was not collected for any participants. Because of the bias in who qualified for the study it became apparent we would not get any statistically valid results.
Arm/Group | Wavefront Optimized LASIK | Wavefront Optimized Photorefractive Keratectomy | Topography-guided LASIK | Topography-guided Photorefractive Keratectomy
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Change in Contrast Sensitivity From Baseline to Month 3
Description: Contrast sensitivity will be tested pre-operatively and 3 months post-operatively
Time Frame: 3 months
Population: Per 2018 protocol amendment contrast sensitivity assessment was removed from the study procedures and thus data was not collected.
Arm/Group | Wavefront Optimized LASIK | Wavefront Optimized Photorefractive Keratectomy | Topography-guided LASIK | Topography-guided Photorefractive Keratectomy
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Other Pre Specified Outcome: Change in Quality of Life Score From Baseline to 3 Months
Description: The validated Quality of Life Impact of Refractive Correction survey will be administered pre-operatively and 3 months post surgery
Time Frame: 3 months
Population: The Quality of Life Impact of Refractive Correction survey was removed from the protocol with the 2018 amendment, thus this data was not collected.
Arm/Group | Wavefront Optimized LASIK | Wavefront Optimized Photorefractive Keratectomy | Topography-guided LASIK | Topography-guided Photorefractive Keratectomy
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Wavefront Optimized LASIK | Wavefront Optimized Photorefractive Keratectomy | Topography-guided LASIK | Topography-guided Photorefractive Keratectomy
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/20 | 0/18 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/20 | 0/18 | 0/20
Other Adverse Events (participants affected / at risk) | 0/18 | 0/20 | 0/18 | 0/20

LIMITATIONS AND CAVEATS:
The study was terminated early. Because of strong selection bias in who qualified for the study, it became apparent we would not get any statistically valid results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/76/NCT03075176/Prot_SAP_001.pdf